CLINICAL TRIAL: NCT04997317
Title: Treatment of Recurrent or Progressive Meningiomas With the Radiolabelled Somatostatin Antagonist 177Lu-Satoreotide (PROMENADE-Study)
Brief Title: Treatment of Recurrent or Progressive Meningiomas With the Radiolabelled Somatostatin Antagonist 177Lu-satoreotide
Acronym: PROMENADE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Cancer League (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00303; th21Wild2
Record Dates: First submitted 2021-07-19; First posted 2021-08-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Meningioma
Keywords: tumour; intercranial neoplasms; peptide receptor radionuclide therapy (PRRT); radiolabelled somatostatin antagonists; cancer; somatostatin receptors; 177Lu-DOTA-JR11; 77Lu-DOTATOC; somatostatin receptor subtype 2 (sstr2); 177Lu-satoreotide
MeSH Terms: conditions — Meningioma; Neoplasms | interventions — 177Lu-DOTA-JR11; Crossing Over, Genetic; 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Intervention Model Description: This is a, two-step, cross-over, open-label phase 0 study comparing the therapeutic index of 177Lu-DOTA-JR11 and 177Lu-DOTATOC followed by a single-arm open-label Phase I/II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 0: Group A (Active Comparator): Cycle 1: 4.5 GBq 177Lu-DOTA-JR11 (300-1300 μg) will be administered once intravenously.
  Cycle 2: 4.5 GBq 177Lu-DOTATOC (≈200 μg) will be administered once intravenously (following a cross-over design).
  Cycle 3 and Cycle 4 will be performed for group A patients with 7.4 GBq 177Lu-DOTATOC (clinically established amount of activity). Cycle 3 and 4 are standard of care (i.e. not part of the study).
  Interventions: Drug: 177Lu-DOTA-JR11 (Phase 0); Cycle 1 and Cycle 2 (cross-over); Drug: 177Lu-DOTATOC (Phase 0); Cycle 1 and Cycle 2 (cross-over), Cycle 3 and 4
- Phase 0: Group B (Active Comparator): Cycle 1: 4.5 GBq 177Lu-DOTATOC (≈200 μg) will be administered once intravenously.
  Cycle 2: 4.5 GBq 177Lu-DOTA-JR11 (300-1300 μg) will be administered once intravenously (following a cross-over design).
  Cycle 3 and Cycle 4 will be performed for group B patients with 7.4 GBq 177Lu-DOTATOC (clinically established amount of activity). Cycle 3 and 4 are standard of care (i.e. not part of the study).
  Interventions: Drug: 177Lu-DOTA-JR11 (Phase 0); Cycle 1 and Cycle 2 (cross-over); Drug: 177Lu-DOTATOC (Phase 0); Cycle 1 and Cycle 2 (cross-over), Cycle 3 and 4
- Phase I/II (Active Comparator): 3 cycles of 177Lu-DOTA-JR11 will be administered with an activity of 4.5-7.4 GBq. Two additional 177Lu-DOTA-JR11 treatment cycles can be performed if clinically indicated
  Interventions: Drug: 177Lu-DOTA-JR11 (Phase I/II)

INTERVENTIONS:
Drug: 177Lu-DOTA-JR11 (Phase 0); Cycle 1 and Cycle 2 (cross-over) — 177Lu-DOTA-JR11 has three main components, namely the somatostatin analogue JR11, the chemical chelator group DOTA and the beta emitter 177Lutetium (177Lu). In the Phase 0 part of the study 177Lu-DOTA-JR11 will be administered once intravenously. The activity of the first 2 cycles will be capped at 4.5 GBq (range: 4.2-4.6 GBq).
  Arms: Phase 0: Group A; Phase 0: Group B
Drug: 177Lu-DOTATOC (Phase 0); Cycle 1 and Cycle 2 (cross-over), Cycle 3 and 4 — 177Lu-DOTATOC is a therapeutic medicinal product and has 3 main components (a) 177Lutetium (177Lu), a beta-emitting radionuclide with a half-life of 6.64 days; (b) DOTA, a chemical chelator group; and (c) TOC (= [Tyr]3-octreotide) an agonistic somatostatin analogue which binds to sstr2 and sstr5 receptors. In the Phase 0 part of the study 177Lu-DOTATOC will be administered once intravenously. The activity of the first 2 cycles will be capped at 4.5 GBq (range: 4.2-4.6 GBq). The remaining 2 cycles will be performed with an activity of 7.4 GBq 177Lu-DOTATOC (total number of cycles = 4).
  Arms: Phase 0: Group A; Phase 0: Group B
Drug: 177Lu-DOTA-JR11 (Phase I/II) — In the phase I/II part of the study: 3 cycles of 177Lu-DOTA-JR11 will be administered with an activity of 4.5-7.4 GBq. Two additional 177Lu-DOTA-JR11 treatment cycles can be performed if clinically indicated
  Arms: Phase I/II

SUMMARY:
Meningiomas are known to be the most frequent intracranial neoplasms and account for approx. 25-33% of all intracranial tumours.Targeted radionuclide therapy with radiolabelled somatostatin analogues, also called Peptide Receptor Radionuclide Therapy (PRRT), has proven to be an effective treatment in metastatic intestinal neuroendocrine tumours and is currently used in advanced, recurrent or progressive meningiomas with promising results. In this study, the therapeutic index of a standard and newly developed radiolabelled somatostatin antagonist will be evaluated and compared in PRRT. In a second step, safety and efficacy of the latter will be assessed.

DETAILED DESCRIPTION:
The somatostatin receptor subtype 2 (sstr2) has been identifies as a peptide hormone receptor that is highly expressed in 70 - 100% of meningiomas representing an attractive target for so called "theranostic" applications combining molecular imaging and targeted radionuclide therapy with radiolabelled somatostatin analogues.The newly developed radiolabelled somatostatin antagonist 177Lu-DOTA-JR11 has been shown to exert a high binding affinity to sstr2 suggesting a higher efficacy in the treatment of advanced meningiomas than the currently available somatostatin analogues (e.g. 177Lu-DOTATOC, 177Lu-DOTATATE).Therefore, the hypothesis has been postulated that 177LuDOTA-JR11 has an improved therapeutic index (tumour-to-dose limiting organ dose ratios) compared to 177Lu-DOTATOC, and that it can be safely used for PRRT in patients with advanced, recurrent or progressive meningiomas. The aim of this 2-step Phase 0 / Phase I/II study is to a) evaluate in the same meningioma patients the therapeutic index (tumour-to-dose limiting organ dose ratios) of 177Lu-DOTA-JR11 in comparison to 177Lu-DOTATOC and b) based on the previous results, to evaluate safety and preliminary efficacy of PRRT with 177Lu-DOTA-JR11.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Participants of any gender and of age > 18 years
* Female participants capable of giving birth (who are not surgically sterilized or are less than 2 years in their menopause) must use a medically accepted contraceptive and must agree to use it during and till 3 months after the treatment. As acceptable contraceptive count sexual abstinence or double contraceptive methods: hormonal contraceptive (oral, transdermal, implants or injections) in combination with barrier methods (spiral, condom, diaphragm)
* Male participants must use medically accepted contraceptive during and till 3 months after treatment
* The participants' Karnofsky Performance Status must be ≥ 60
* The participants must be patients with a histologically or clinically confirmed (MRI + somatostatin receptor imaging) recurrent or progressive meningioma
* There must be no other standard therapeutic alternatives for the participants
* The participants tumour must be measurable according to RECIST v1.1 with a minimal diameter of 1.0 cm.
* The participants must have a confirmed expression of somatostatin receptor (SSTR) on 68Ga- DOTATOC positron emission computed tomography (PET)/CT scan
* Blood parameter criteria are:

  h) Leucocytes ≥ 3*109/L i) Haemoglobin ≥ 80 g/L j) Thrombocytes ≥ 90*109/L k) Estimated glomerular filtration rate ≥ 50 ml/min l) Albumin > 25g/L m) alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (AP): ≤ 5 times upper standard value n) Bilirubin ≤ 2 times upper standard value

Exclusion Criteria:

* Known intolerance against 177Lu, DOTA, JR11, TOC or against one of the components of 177Lu-DOTA-JR11 or 177Lu-DOTATOC
* Ongoing infection at the screening visit or a serious infection in the past 4 weeks
* Administration of another investigational product in the last 60 days before Visit 1 Day 1
* Prior or planed administration of a therapeutic radio-pharmaceutical during 8 half-lives of the used radio-pharmaceutical's radionuclide, also during the ongoing study
* Any extensive Radiotherapy involving bone marrow over the last 3 months before inclusion to the study
* Chemotherapy in the last 2 months before inclusion
* Pregnant or breastfeeding female patients. A pregnancy test will be performed in all women of child bearing potential.
* Any uncontrolled significant medical, psychiatric or surgical condition (active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus [HbA1c ≥ 9%], uncontrolled congestive heart disease, etc.) or laboratory findings that might jeopardize the patient's safety or that would limit compliance with the objectives and assessments of the study. Any mental conditions which prevent the patient from understanding the type, extent and possible consequences of the study and/or an uncooperative attitude from the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Tumour-to-dose limiting organ dose ratio T-to-bone marrow: Therapeutic Index (Phase 0) | 24, 48 and 168 hours (+/- 30 min up to 24 hours)
  Radiation Dosimetry of the Radiopharmaceuticals 177Lu-DOTA-JR11 and 177Lu-DOTATOC. In Phase 0 the primary objective is to assess the tumour-to-bone marrow dose ratios of 177Lu-DOTA-JR11 and 177Lu-DOTATOC. In order to get kinetic information of 177Lu- DOTA-JR11 and 177Lu-DOTATOC for this task total body scintigraphy and SPECT/CT of head and abdomen (phase 0 study) or only head (phase I/II study) are performed at different time points post injection 177Lu-DOTA-JR11 or 177Lu-DOTATOC.
Change in Tumour-to-dose limiting organ dose ratio T-to-kidney: Therapeutic Index (Phase 0) | 24, 48 and 168 hours (+/- 30 min up to 24 hours)
  Radiation Dosimetry of the Radiopharmaceuticals 177Lu-DOTA-JR11 and 177Lu-DOTATOC. In Phase 0 the primary objective is to assess the tumour-to-kidney dose ratios of 177Lu-DOTA-JR11 and 177Lu-DOTATOC. In order to get kinetic information of 177Lu- DOTA-JR11 and 177Lu-DOTATOC for this task total body scintigraphy and SPECT/CT of head and abdomen (phase 0 study) or only head (phase I/II study) are performed at different time points post injection 177Lu-DOTA-JR11 or 177Lu-DOTATOC.
Assessment of treatment safety (phase I/II) by number of AEs graded according to CTCAE v5.0 | About 1 hour before infusion up to 41 - 45 days after infusion
  In Phase I/II the primary objective is to assess the safety considerations of patients treated with 177Lu-DOTA-JR11 after 3 - 5 cycles of 177Lu-DOTA-JR11 PRRT: AEs graded according to CTCAE v5.0

SECONDARY OUTCOMES:
Tumour absorbed dose (Gy) (Phase 0 and phase I/II) | up to 40 weeks
  Assessment of maximal tumour absorbed dose (Gy) and dose coefficient (mGy/MBq) (two first cycles only)
Organ absorbed dose (Gy) (Phase 0) | up to 40 weeks
  Assessment of organ absorbed dose (Gy) and dose coefficient (mGy(MBq) (two first cycles only)
Organ and tumour residence time (Phase 0) | up to 40 weeks
  Assessment of organ and tumour residence time (time integrated activity coefficient) (two first cycles only)
Tumour-to-remaining organ dose ratio (Phase 0) | up to 40 weeks
  Assessment of tumour-to-remaining organ dose ratios (not dose limiting organs, e.g. tumour-to-spleen) (two first cycles only)
Evaluation radiation doses (Phase 0 and Phase II) | up to 40 weeks
  Assessment and comparison of whole body and organ radiation doses of 177Lu-DOTA-JR11 (first cycle only)
Early onset toxicity (Phase 0) | up to 20 weeks
  Assessment of safety (early onset toxicity): Adverse events (AEs) graded according to CTCAE v5.0 (two first cycles only)
Change in Quality of life (QoL) short form (SF) 36 questionnaire (Phase 0 and I/II) | From Screening up to 12 months after 3rd infusion
  Assessment of QoL SF36 questionnaire: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Change in visual parameters (Phase 0 and Phase I/II) | up to 60-70 weeks
  For optical nerve sheath meningiomas: Assessment of visual acuity (visual field) before and after start with PRRT.
Change in Plasma Concentration [Cmax] of 177Lu-DOTA-JR11 in the human body (Phase I/II) | up to 50 weeks
  Assessment of pharmacokinetics of 177Lu-DOTA-JR11 in the human body.
Whole body and organ radiation doses (Phase I/II) | up to 60-70 weeks
  Assessment of whole body and organ radiation doses of 177Lu-DOTA-JR11 (first cycle only)

OTHER OUTCOMES:
Assessement of Progression-Free Survival (PFS) (Phase 0 and I/II)) | up to 12 months
  PFS rate will be evaluated by MRI 6 and 12 months after start with first treatment cycle with 177Lu-DOTA-JR11.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Cordier, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Neurosurgery, Basel, Canton of Basel-City, Switzerland